CLINICAL TRIAL: NCT00123409
Title: Telephone Disease Management At-Risk Drinking (TDM 11)
Brief Title: Telephone Disease Management At-Risk Drinking (TDM II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 02-108
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-06

CONDITIONS: Alcohol Abuse
Keywords: Primary Care; Telephone; Quality of Life
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone Disease Management (Experimental): Telephone based disease management or counseling used to promote a reducution in alcohol misuse
  Interventions: Behavioral: Telephone disease management
- Usual Care (Placebo Comparator): Usual Care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Telephone disease management — Telephone based care management
  Arms: Telephone Disease Management
Behavioral: Usual Care — Usual care
  Arms: Usual Care

SUMMARY:
The aim of this study is to test for improvements in treatment outcomes for primary care patients with at-risk drinking when cared for using telephone disease management (TDM) compared to those treated with usual care. Based on our pilot data, TDM for at-risk drinking may be a viable method for reducing alcohol consumption in this population.

Hypotheses: The hypotheses for this research plan are: 1. A significantly greater proportion of patients assigned to TDM will obtain improvement in drinking outcomes compared to usual care. 2. TDM will lead to greater access to behavioral health care and higher intensity of treatment relative to usual care. This effect will be moderated by logistics such as transportation problems, physical functioning, and employment status. 3. More patients assigned to TDM will receive guideline adherent care.

DETAILED DESCRIPTION:
We propose to randomize 200 patients with at-risk drinking from four primary care clinics at the PVAMC and three Community Based Outpatient Clinics (CBOCs). Patients will be identified for participation by 1. referrals from primary care clinicians based on existing screening and clinical exams or 2. from the screening of a random subset of patients with an appointment in the primary care clinic. A baseline assessment will establish eligibility for participation in the study. The baseline assessment will also allow identification of those patients who screen positive but do not have a definable behavioral health problem and those with severe symptoms who may need more intensive help than provided by the study.

Consenting eligible patients will be randomly assigned to TDM or the lower intensity intervention of usual care. For those patients assigned to usual care, the physician will administer further evaluations and treatment as he/she sees fit. For those assigned to TDM, the primary care provider remains the agent of treatment, but a Behavioral Health Specialist (BHS) is made available to: maintain regularly scheduled telephone contact, develop a treatment plan, monitor treatment effectiveness, assess and encourage treatment adherence, and offer support and education. The role of the health specialist is defined by a treatment manual that adheres to the recommendations of VA practice guidelines. TDM is based on a chronic care model of treatment and includes a minimum of three BAI sessions. The health specialist will communicate assessment information with the PCP in order to coordinate treatment decisions.

The principal outcomes of the study relate to reduction in alcohol use within recommended guidelines as well as access and utilization of behavioral health services over the course of 12 months. Results favoring TDM may provide a low-cost, highly efficient mechanism for integrating behavioral health with primary care for these patients. This project thus meets several of the priority areas for HSR&D funding including improving access to care, the implementation of practice guidelines, use of telemedicine, and patient-centered care.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years of age and over, male or female.
* meet criteria for at-risk drinking as defined by drinking more than 21 standard drinks per week (14 for women or those over age 65).

Exclusion Criteria:

* show an absence of any of the following:

  1. active suicidal ideation,
  2. regular current use of illicit substances other than alcohol
  3. diagnosis of current alcohol dependence
  4. current hallucinations and delusions
  5. current symptoms of PTSD
  6. a history of mania or hypomania.
* have adequate hearing to participate in telephone assessments and access to a telephone. Subjects will also show an absence of other barriers to verbal communication (e.g., aphasia) and will be cognitively intact (Brief Orientation Memory and Concentration task greater than 15 for those over age 54).
* not actively participating in specialized addiction treatment within the prior 3-months.
* not currently enrolled in another clinical trial
* not expected to move from the VISN 4 area within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2004-01; Primary Completion 2008-08 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W. Oslin, MD, Principal Investigator — Philadelphia VA Medical Center, Philadelphia, PA
Locations (1):
- Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Datto CJ, Thompson R, Horowitz D, Disbot M, Oslin DW. The pilot study of a telephone disease management program for depression. Gen Hosp Psychiatry. 2003 May-Jun;25(3):169-77. doi: 10.1016/s0163-8343(03)00019-7. PMID 12748029
- [Result] Oslin DW, Ross J, Sayers S, Murphy J, Kane V, Katz IR. Screening, assessment, and management of depression in VA primary care clinics. The Behavioral Health Laboratory. J Gen Intern Med. 2006 Jan;21(1):46-50. doi: 10.1111/j.1525-1497.2005.0267.x. PMID 16423122
- [Result] Oslin DW, Sayers S, Ross J, Kane V, Ten Have T, Conigliaro J, Cornelius J. Disease management for depression and at-risk drinking via telephone in an older population of veterans. Psychosom Med. 2003 Nov-Dec;65(6):931-7. doi: 10.1097/01.psy.0000097335.35776.fb. PMID 14645769
- [Result] McKay JR, Van Horn DH, Oslin DW, Lynch KG, Ivey M, Ward K, Drapkin ML, Becher JR, Coviello DM. A randomized trial of extended telephone-based continuing care for alcohol dependence: within-treatment substance use outcomes. J Consult Clin Psychol. 2010 Dec;78(6):912-23. doi: 10.1037/a0020700. PMID 20873894
- [Result] McKay JR, Van Horn D, Oslin DW, Ivey M, Drapkin ML, Coviello DM, Yu Q, Lynch KG. Extended telephone-based continuing care for alcohol dependence: 24-month outcomes and subgroup analyses. Addiction. 2011 Oct;106(10):1760-9. doi: 10.1111/j.1360-0443.2011.03483.x. Epub 2011 Aug 8. PMID 21545667

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Telephone Based care management for reducing alcohol use
  Telephone disease management: Telephone based care management
- Arm 2: Usual Care
  Usual Care: Usual care
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 72 | 74
Completed | 68 | 71
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Telephone Disease Management: Telephone Based care management for reducing alcohol use
  Telephone disease management: Telephone based care management
- Total: Total of all reporting groups
Arm/Group | Telephone Disease Management | Usual Care | Total
Number analyzed (Participants) | 68 | 71 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (15.1) | 57 (13.9) | 57.1 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 67 | 69 | 136
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 33 | 63
  White | 38 | 38 | 76
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 68 | 71 | 139
# of Days Drinking in last 28 days [Mean (Standard Deviation); unit: # of days drinking] | 19.53 (9.44) | 20.2 (8.12) | 19.9 (8.8)
Problems related to alcohol [Mean (Standard Deviation); unit: # problems] — Measure used was the Short Inventory of Problem Drinking (SIP)
  # problems | 4.31 (5.52) | 4.7 (5.52) | 4.5 (5.52)

OUTCOME MEASURES:

1. Primary Outcome: Reduced Alcohol Use
Description: Alcohol use as measured by the number of drinking days. Lower is better. There are no upper limits. The lower limit is 0.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Days drinking
Groups:
- Telephone Based Management: Telephone Based Management used to reduce alcohol misuse
  Telephone disease management: Telephone based care management
Arm/Group | Telephone Based Management | Usual Care
Number analyzed (Participants) | 68 | 71
Days drinking | 14.96 (12.55) | 15.52 (10.12)

2. Secondary Outcome: Reduced Problems Related to Alcohol
Description: The Short Inventory of Problmes was used to measure the number of alcohol related problems encountered in the prior 3 months. The scale has a minimum of 0 with lower as better. The max score is 15 with each problem rated as present or absent.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: # of alcohol problems
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 68 | 71
# of alcohol problems | 2.37 (5.11) | 2.77 (6.24)

ADVERSE EVENTS:
Time Frame: the 12 months of the intervention
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/71
Other Adverse Events (participants affected / at risk) | 0/68 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No